CLINICAL TRIAL: NCT01813383
Title: Clinical Relevance of Typing HLA-DR7-DQ2
Acronym: HLA
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Juan Francisco Delgado de la Poza, Medicine. Immunology specialist, Corporacion Parc Tauli
Other Study IDs: Celiac disease and HLA-DQ2.2
Record Dates: First submitted 2013-03-12; First posted 2013-03-19 (Estimated); Last update posted 2013-03-19 (Estimated); Status verified 2013-03

CONDITIONS: Celiac Disease Patients Following Recommendations of ESPGHAN; HLA-DQ2 Typing Include HLA-DR7-DQ2 Haplotypes
Keywords: Celiac disease; HLA-DQ2.2; HLA-DQ2.5; HLA-DR7-DQ2; HLA-DR3-DQ2
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- HLA-DR3-DQ2 patients: Patients with HLA-DR3-DQ2 haplotype
  Interventions: Other: There is not any intervention
- HLA-DR7-DQ2 patients: Patients with HLA-DR7-DQ2 haplotype
  Interventions: Other: There is not any intervention

INTERVENTIONS:
Other: There is not any intervention

SUMMARY:
Celiac disease patients with HLA-DR7-DQ2 haplotype have the same histological, analytical and clinical behaviour as patients with HLA-DR3-DQ2 haplotype.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of celiac disease following ESPGHAN recommendations
* HLA-DQ2 typing including HLA-DR3-DQ2 and HLA-DR7-DQ2 haplotypes

Exclusion Criteria:

* Patients who have not been diagnosed for celiac disease
* HLA-DQ2 typing that not include HLA-DR7-DQ2 haplotype

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Celiac disease patients who have been diagnosed in a Hospital by a Pediatrician.
Sampling Method: Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Anti-tissue transglutaminase | Up to 1 month after diagnosis

SECONDARY OUTCOMES:
Anti-Endomysium autoantibodies | Up to 1 month after diagnosis

OTHER OUTCOMES:
Oberhuber histological damage classification | Up to 1 month after diagnosis
Clinical characteristics of celiac disease | Up to 1 month after diagnosis
  Asymptomatic, intestinal symptoms, extra-intestinal symptoms, European Society for Pediatric Gastroenterology, Hepatology, and Nutrition (ESPGHAN) score

CONTACTS AND LOCATIONS:
Overall Officials: Juan Francisco Delgado de la Poza, Principal Investigator — Immunology Section, Laboratori. UDIAT-CD. Corporació Sanitària i Universitària Parc Taulí
Locations (1):
- Corporació Sanitària i Universitària Parc Taulí, Sabadell, Barcelona, Spain